CLINICAL TRIAL: NCT00394654
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Evaluate the Efficacy of MEDI-528, a Humanized Anti-Interleukin-9 Monoclonal Antibody, on Late Asthmatic Response Induced By Allergen Inhalation In Adults With Atopic Asthma
Brief Title: A Study to Evaluate the Efficacy of MEDI-528 on Late Asthmatic Response With Atopic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP138; NCT00394654 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — enokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDI528 9 mg/kg (Experimental): MEDI-528 at a single dose of 9 mg/kg administered as an intravenous infusion
  Interventions: Biological: MEDI-528 9 mg/kg
- PLACEBO (Placebo Comparator): Placebo administered as a single intravenous infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI-528 9 mg/kg — MEDI-528 at a single dose of 9 mg/kg administered as an intravenous infusion
  Arms: MEDI528 9 mg/kg
Other: Placebo — Placebo administered as a single intravenous infusion
  Arms: PLACEBO

SUMMARY:
This is a Phase 2a, randomized multicenter study to evaluate the efficacy of MEDI-528 on LAR in adult patients with atopic asthma.

DETAILED DESCRIPTION:
This study (MI-CP138) is a Phase 2a, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy of MEDI-528 on LAR in adult patients with atopic asthma. Approximately three investigative sites in Canada will participate in this study, with up to 40 evaluable patients randomized in a 1:1 ratio to receive MEDI-528 (9.0 mg/kg) or placebo as a single IV infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, age 18 through 65 years of age at the time of screening;
* Written informed consent obtained from the patient prior to receipt of any study medication or beginning study procedures;
* Previously documented diagnosis of asthma of > 1 year duration, based on episodic symptoms of airflow obstruction, at least partial reversibility of airflow obstruction, with alternative diagnoses (e.g., chronic obstructive pulmonary disease) ruled out;
* AHR in the methacholine challenge test with a PC20 (provoking concentration of methacholine to cause a 20% fall in FEV1) ≤ 16 mg/mL (Crapo, 2000);
* Have dual response of EAR, defined as a decrease in FEV1 ≥ 20% at 0 to 3 hours after inhalation, and LAR, defined as a decrease in FEV1 ≥ 15% 3 to 7 hours after inhalation, to inhaled allergen;
* Asthma symptoms are adequately controlled on short-acting β2 agonists (e.g., albuterol) alone;
* Have had no significant changes in regular asthma medications and no acute asthma exacerbations requiring corticosteroid rescue, hospitalization, or emergency department visits for at least 4 weeks prior to screening and up through the time of the first dose of study drug on Study Day 0.
* Sexually active women, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 21 days prior to the first dose of study drug on Study Day 0, and must agree to continue using such precautions through Study Day 126. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active men, unless surgically sterile, must likewise use an effective method of birth control (condom) and must agree to continue using such precautions through Study Day 126;
* Able to complete the follow-up period through Study Day 126, as required by the protocol.
* Willing to forego other forms of experimental treatment and study procedures during the study; and
* Able to provide spirometric readings that meet American Thoracic Society (ATS) standards (ATS, 1995).

Exclusion Criteria:

* Receipt of MEDI-528 in any previous clinical study;
* History of allergy or adverse reactions to any component of the MEDI-528 formulation;
* Lung disease other than allergic asthma (e.g. chronic bronchitis);
* Current use of any systemic or inhaled immunosuppressive drugs, including systemic and inhaled corticosteroids (topical corticosteroids are permitted), long-acting β2 agonists, leukotriene antagonists, cromolyn sodium, nedocromil sodium, theophylline or any inhaled or systemic medication for asthma other than short-acting β2 agonists, for at least 4 weeks prior to study drug administration on Study Day 0.
* Current use of any β-adrenergic antagonist (e.g. propranolol).
* Any disease or illness, other than asthma, that may require the use of systemic corticosteroids during the study period.
* Acute illnesses or evidence of clinically significant active infection, such as fever ³ 38.0°C (100.5°F) at screening and through the time of the study drug administration on Study Day 0;
* Current allergy-vaccination therapy (i.e., desensitization immunotherapy) with less than 3 months of stable maintenance doses prior to the baseline allergen inhalation challenge;
* Receipt of any investigational drug therapy within 30 days or any biologic(s) within 5 half-lives of the agent prior to the first dose of study drug through Study Day 150;
* Receipt of any therapy with a leukocyte-depleting agent unless recovery in white cell count has been documented before screening;
* Pregnancy (sexually active females must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to study drug administration on Study Day 0);
* Is a nursing mother at the time of study enrollment;
* Evidence of infection with hepatitis B or C virus, or HIV-1 or HIV-2, or active infection with hepatitis A;
* History of significant systemic disease (e.g., cancer; infection; coronary artery disease or other cardiovascular disease; or hematological, renal, hepatic, endocrinologic, neurologic, rheumatologic, or gastrointestinal disease);
* History of cancer other than nonmelanoma skin cancer or cervical carcinoma-in-situ that have been treated successfully with curative therapy;
* History of primary immunodeficiency;
* History of pancreatitis;
* History of use of tobacco products within 2 years of baseline or history of smoking >= 10 pack-years;
* Elective surgery planned from the time of screening through Study Day 126;
* Clinically significant abnormalities (other than asthma) upon physical examination prior to study drug administration on Study Day 0;
* Clinically significant abnormality, as determined by the investigator, on 12-lead ECG or chest radiograph at the time of screening;
* At the time of screening, any of the following abnormalities: aspartate transaminase (AST), alanine transaminase (ALT), or amylase > 1.5 × above the upper limits of normal (ULN); or serum creatinine > 1.3 × ULN; or any other abnormal laboratory values in the screening panel that, in the opinion of the principal investigator (PI), are judged to be clinically significant; or
* Evidence of any systemic disease or respiratory disease (other than asthma), any finding upon physical examination or history of any disease that, in the opinion of the PI or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Molfino, M.D., Study Director — MedImmune LLC
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Hopital Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty patients were entered into the study between 16Oct2006 and 15Aug2007 at 2 sites in Canada.
Pre-assignment Details: Treatment assignments were determined using a block randomization procedure with a 1:1 ratio through an interactive Web response system (IWRS). Patients who were randomized into the study but did not complete the second allergen challenge on Day 7 were replaced, unless the patient withdrew for safety reasons.
Groups:
- MEDI528 9 mg/kg: MEDI-528 at a single dose of 9 mg/kg administered as an IV infusion
Period: Overall Study
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Started | 15 | 15
Completed | 13 | 15
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — PARTICIPANT LEFT STDUY REGION | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | MEDI528 9 mg/kg | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (9.6) | 26.5 (7.8) | 28.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Effect of MEDI-528 on Late Asthmatic Response (LAR) After Inhaled Allergen Challenge at Day 7
Description: Change from baseline (percent reduction) in mean maximum decline of forced expiratory volume in one second (FEV1) during LAR at 3 to 7 hours after an inhaled allergen challenge.
Time Frame: Day 7
Population: All participants who were randomized into the study and completed the second allergen challenge on Day 7.
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- PLACEBO: Placebo administered as a single intravenous (IV) infusion
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 13 | 12
Percent | 21.26 (69.288) | -16.21 (61.788)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 9 mg/kg; Test type: Superiority or Other; p = 0.168, Univariate 2-sample t-test

2. Primary Outcome: Effect of MEDI-528 on LAR After Inhaled Allergen Challenge at Day 28
Description: Change from baseline (percent reduction) in mean maximum decline of FEV1 during LAR at 3 to 7 hours after an inhaled allergen challenge.
Time Frame: Day 28
Population: All participants who were randomized into the study and completed the second allergen challenge on Day 7.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 14 | 11
Percent | 29.93 (46.646) | -16.95 (123.256)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 9 mg/kg; Test type: Superiority or Other; p = 0.254, Univariate 2-sample t-test

3. Primary Outcome: Effect of MEDI-528 on LAR After Inhaled Allergen Challenge at Day 56
Description: as for outcome 2
Time Frame: Day 56
Population: All participants who were randomized into the study and completed the second allergen challenge on Day 7.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 13 | 11
Percent | 40.36 (45.123) | 31.85 (53.709)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 9 mg/kg; Test type: Superiority or Other; p = 0.677, Univariate 2-sample t-test

4. Primary Outcome: Effect of MEDI-528 on LAR After Inhaled Allergen Challenge at Day 7
Description: Change from baseline (percent reduction) in mean maximum decline of area under the concentration-time curve (AUC) of the participants FEV1 during LAR at 3 to 7 hours after an inhaled allergen challenge.
Time Frame: Day 7
Population: All participants who were randomized into the study and completed the second allergen challenge on Day 7.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 13 | 12
Percent | 21.86 (94.34) | -14.47 (82.43)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 9 mg/kg; Test type: Superiority or Other; p = 0.318, Univariate 2-sample t-test

5. Primary Outcome: Effect of MEDI-528 on LAR After Inhaled Allergen Challenge at Day 28
Description: Change from baseline (percent reduction) in mean maximum decline of AUC of the participants FEV1 during LAR at 3 to 7 hours after an inhaled allergen challenge.
Time Frame: Day 28
Population: All participants who were randomized into the study and completed the second allergen challenge on Day 7.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 14 | 11
Percent | 2.91 (133.75) | -13.09 (175.27)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 9 mg/kg; Test type: Superiority or Other; p = 0.798, Univariate 2-sample t-test

6. Primary Outcome: Effect of MEDI-528 on LAR After Inhaled Allergen Challenge at Day 56
Description: as for outcome 5
Time Frame: Day 56
Population: All participants who were randomized into the study and completed the second allergen challenge on Day 7.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 13 | 11
Percent | 41.75 (65.49) | 51.91 (98.49)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 9 mg/kg; Test type: Superiority or Other; p = 0.766, Univariate 2-sample t-test

7. Secondary Outcome: Incidence of Adverse Events
Description: Number of participants experiencing adverse events (includes both adverse events and serious adverse events)
Time Frame: Days 0 - 126
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 15 | 15
Participants | 11 | 12

8. Secondary Outcome: Incidence of Serious Adverse Events
Description: Number of participants experiencing serious adverse events
Time Frame: Days 0 - 126
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 15 | 15
Participants | 1 | 0

9. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) to MEDI-528
Description: Number of participants with ADA to MEDI-528
Time Frame: Days 0, 27, 55, 84, and 126
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

10. Secondary Outcome: Time to Observed Maximum Serum Concentration (Tmax)
Description: Tmax of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Day |  | 0.028 (20.4)

11. Secondary Outcome: Time to Observed Maximum Sputum Concentration (Tmax)
Description: Tmax of MEDI-528 in sputum
Time Frame: Days -21 to -7, 7, 28, and 56
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Day |  | 9.276 (99)

12. Secondary Outcome: Time to Observed Maximum Nasal Lavage Concentration (Tmax)
Description: Tmax of MEDI-528 in nasal lavage
Time Frame: Days -6 to -1, 8, 29, and 57
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Day |  | 10.319 (169.6)

13. Secondary Outcome: Observed Maximum Serum Concentration (Cmax)
Description: Cmax of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Microgram per milliliter |  | 229.672 (18.1)

14. Secondary Outcome: Observed Maximum Sputum Concentration (Cmax)
Description: Cmax of MEDI-528 in sputum
Time Frame: Days -21 to -7, 7, 28, and 56
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Nanogram per milliliter |  | 71.843 (78.7)

15. Secondary Outcome: Observed Maximum Nasal Lavage Concentration (Cmax)
Description: Cmax of MEDI-528 in nasal lavage
Time Frame: Days -6 to -1, 8, 29, and 57
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Nanogram per milliliter |  | 79.406 (136.6)

16. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Last Measurable Concentration [AUC(0-t)]
Description: AUC(0-t) of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Microgram times day per milliliter |  | 5744.821 (14.8)

17. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Last Measurable Concentration [AUC(0-t)]
Description: AUC(0-t) of MEDI-528 in sputum
Time Frame: Days -21 to -7, 7, 28, and 56
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Nanogram times day per milliliter |  | 2382.123 (84)

18. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Last Measurable Concentration [AUC(0-t)]
Description: AUC(0-t) of MEDI-528 in nasal lavage
Time Frame: Days -6 to -1, 8, 29, and 57
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Nanogram times day per milliliter |  | 1332.408 (147.6)

19. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Infinity [AUC(0-infinity)]
Description: AUC(0-infinity) of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Microgram times day per milliliter |  | 6224.272 (17)

20. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Infinity [AUC(0-infinity)]
Description: AUC(0-infinity) of MEDI-528 in sputum
Time Frame: Days -21 to -7, 7, 28, and 56
Population: All participants who were randomized, received any MEDI-528, and had sputum samples obtained
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 10
Nanogram times day per milliliter |  | 4136.234 (61.9)

21. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Infinity [AUC(0-infinity)]
Description: AUC(0-infinity) of MEDI-528 in nasal lavage
Time Frame: Days -6 to -1, 8, 29, and 57
Population: All participants who were randomized, received any MEDI-528, and had nasal lavage samples obtained
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 10
Nanogram times day per milliliter |  | 6047.098 (134)

22. Secondary Outcome: Percent of Total Area Under the Concentration Curve Extrapolated From Last Measurable Time to Infinity [AUC(Ext)]
Description: AUC(ext) of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Percent |  | 6.441 (59.3)

23. Secondary Outcome: Percent of Total Area Under the Concentration Curve Extrapolated From Last Measurable Time to Infinity [AUC(Ext)]
Description: AUC(ext) of MEDI-528 in sputum
Time Frame: Days -21 to -7, 7, 28, and 56
Population: All participants who were randomized, received any MEDI-528, and had sputum samples obtained
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 10
Percent |  | 25.919 (81.3)

24. Secondary Outcome: Percent of Total Area Under the Concentration Curve Extrapolated From Last Measurable Time to Infinity [AUC(Ext)]
Description: AUC(ext) of MEDI-528 in nasal lavage
Time Frame: Days -6 to -1, 8, 29, and 57
Population: All participants who were randomized, received any MEDI-528, and had nasal lavage samples obtained
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 10
Percent |  | 18.848 (178.3)

25. Secondary Outcome: Terminal Phase Half-Life (T1/2)
Description: T1/2 of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Day |  | 34.316 (20.8)

26. Secondary Outcome: Terminal Phase Half-Life (T1/2)
Description: T1/2 of MEDI-528 in sputum
Time Frame: Days -21 to -7, 7, 28, and 56
Population: All participants who were randomized, received any MEDI-528, and had sputum samples obtained
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 10
Day |  | 31.933 (83.1)

27. Secondary Outcome: Terminal Phase Half-Life (T1/2)
Description: T1/2 of MEDI-528 in nasal lavage
Time Frame: Days -6 to -1, 8, 29, and 57
Population: All participants who were randomized, received any MEDI-528, and had nasal lavage samples obtained
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Day |  | 25.584 (69)

28. Secondary Outcome: Total Body Clearance (CL)
Description: CL of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Liter per day |  | 0.101 (26.7)

29. Secondary Outcome: Terminal Phase Volume of Distribution (Vz)
Description: Vz of MEDI-528 in serum
Time Frame: Days 0, 6, 7, 27, 55, 84, and 126
Population: All participants who were randomized and received any MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 15
Liter |  | 5.025 (23.8)

ADVERSE EVENTS:
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=15) | MEDI528 9 mg/kg (N=15)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=15) | MEDI528 9 mg/kg (N=15)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 4 (6) | 4 (6)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (3)
Lymphocyte count decreased (Investigations) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0)
Protein urine present (Investigations) | 1 (2) | 3 (3)
White blood cell count decreased (Investigations) | 3 (5) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.